CLINICAL TRIAL: NCT01940848
Title: A Double-blind, Randomised, Placebo-controlled Study on the Efficacy of Iberogast® (STW5) in Patients With Irritable Bowel Syndrome
Brief Title: Efficacy/Safety Study to Confirm Iberogast's Efficacy in Patients With Irritable Bowel Syndrome Diagnosed on ROME III Criteria Compared to Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17063; STW5/212-D-011-III-V (Other: Company internal); 2011-002613-10 (EudraCT Number)
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: Iberogast; efficacy; safety
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — iberogast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STW5 (Experimental): 2/3 patients with irritable bowel syndrome will be randomized in this arm
  Interventions: Drug: STW5 (Iberogast, BAY98-7411)
- Placebo (Placebo Comparator): 1/3 patients with irritable bowel syndrome will be randomized in this arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STW5 (Iberogast, BAY98-7411) — Applied orally over 28 days, 20 drops STW 5 three times daily
  Arms: STW5
Drug: Placebo — Applied orally over 28 days, 20 drops placebo three times daily
  Arms: Placebo

SUMMARY:
The study shall prove whether treatment of irritable bowel syndrome with Iberogast is superior to placebo regarding the main criterium "pain"

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged >18 years
* Patients meeting the Rome III irritable bowel syndrome (IBS) diagnostic criteria. IBS is defined as recurrent abdominal pain or discomfort at least 3 days/month in last 3 months (onset at least 6 months ago) associated with two or more of the following:

  * Improvement with defecation
  * Onset associated with a change in frequency of stool
  * Onset associated with a change in form (appearance) of stool
* History of pain intensity with an average of worst abdominal pain in past 24 hours score of > 30 on a daily measured VAS (visual analogue scale) during screening phase

Exclusion Criteria:

* Intake of STW5 within the last 5 years
* Concomitant treatment during the study (including screening phase) with any medication that could influence the gastrointestinal function
* Regular intake of nonsteroidal antiphlogistic drugs incl. COX-2-inhibitors (exception: acetylsalicylic acid for cardiovascular prevention up to 100 mg daily)
* Patients with known hypersensitivity to any component of the trial drugs
* History of eating disorders
* Patients with a history of diseases with abdominal symptoms that can resemble IBS
* Presence of any other acute or chronic gastrointestinal disorder
* History of abdominal surgery (cholecystectomy and appendectomy can be tolerated when performed at least one year previously)
* Known intolerance to azo dyes E 110 and E 151

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2013-10-11 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Number of responders with decrease in pain intensity compared with baseline for at least 14 single days within 4 weeks of treatment | 28 days (+/- 3 days)
  The pain intensity is documented on a 10 cm visual analogue scale (VAS) scale

SECONDARY OUTCOMES:
Number of responders with decrease in pain intensity compared with baseline for at least 7 single days within first 2 weeks of treatment | 14 days (+/- 3 days)
Score on IBS-QOL (Irritable Bowel Syndrome - Quality of Life Measure) scale | 28 days (+/- 3 days)
Stool consistency (IBS-D): Decrease in weekly average of >1 in terms of BSS (Bristol Stool Form Scale) | 28 days (+/- 3 days)
Stool frequency (IBS-C): Increase of 1 or more complete spontaneous bowel movements (CSBM) per week compared with Baseline | 28 days (+/- 3 days)
Numbers of participants with adverse events (AEs) | 28 days (+/- 3 days)
Vital signs | 28 days (+/- 3 days)
  blood pressure, heart rate, body weight
Laboratory parameters | 28 days (+/- 3 days)
  haematology, blood chemistry, urinalysis
Global assessment of tolerability on a 5-point Likert scale by Investigator and patient | 28 days (+/- 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (18):
- Germany (18):
  - Ludwigsburg, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - Sinzheim, Baden-Wurttemberg
  - Potsdam, Brandenburg
  - Lollar, Hesse
  - Wiesbaden, Hesse
  - Wardenburg, Lower Saxony
  - Winsen, Lower Saxony
  - Essen, North Rhine-Westphalia
  - Hagen, North Rhine-Westphalia
  - Löhne, North Rhine-Westphalia
  - Marl, North Rhine-Westphalia
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Halle, Saxony-Anhalt
  - Reinfeld, Schleswig-Holstein
  - Apolda, Thuringia
  - Blankenhain, Thuringia
  - Berlin

REFERENCES:
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/